CLINICAL TRIAL: NCT03102008
Title: An Analysis of Change Processes in the Transdiagnostic Treatment of Emotional Disorders in Adolescents
Brief Title: Unified Protocol for Adolescents (UP-A) Change Processes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Jill May Ehrenreich, Associate Professor, University of Miami
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 20161193
Record Dates: First submitted 2017-03-02; First posted 2017-04-05 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Anxiety Disorders; Depression; Obsessive-Compulsive Disorder; Adolescent - Emotional Problem; Emotional Disorder
Keywords: Transdiagnostic Treatment; Emotional Disorders; Adolescence; Psychotherapy
MeSH Terms: conditions — Anxiety Disorders; Depression; Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of three baseline conditions (2, 3, or 4 week waitlist) and all participants are subsequently treated using the active study intervention (UP-A).
Who Masked: Outcomes Assessor
Masking Description: Independent evaluators to conduct post-treatment evaluations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 2 Week Waitlist (No Intervention): Participants assessed weekly (via self- and parent-report questionnaires administered on the internet) for symptom change during waitlist (baseline) period. At the end of waitlist and prior to treatment phase, symptom/disorder change assessed via clinical interview conducted by independent evaluator.
- 3 Week Waitlist (No Intervention): Participants assessed weekly (via self- and parent-report questionnaires administered on the internet) for symptom change during waitlist (baseline) period. At the end of waitlist and prior to treatment phase, symptom/disorder change assessed via clinical interview conducted by independent evaluator.
- 4 Week Waitlist (No Intervention): Participants assessed weekly (via self- and parent-report questionnaires administered on the internet) for symptom change during waitlist (baseline) period. At the end of waitlist and prior to treatment phase, symptom/disorder change assessed via clinical interview conducted by independent evaluator.
- 16 Sessions of Therapeutic Intervention (Experimental): Participants receive 50 minute sessions weekly of therapeutic intervention (Unified Protocol for the Treatment of Emotional Disorders in Adolescents). Symptom change assessed weekly on the internet or before each session (via self- and parent-report questionnaires). At the end of treatment phase, symptom/disorder change assessed via clinical interview conducted by independent evaluator.
  Interventions: Behavioral: Unified Protocol for Emotional Disorders in Adolescents (UP-A)

INTERVENTIONS:
Behavioral: Unified Protocol for Emotional Disorders in Adolescents (UP-A) — The Unified Protocol for Emotional Disorders in Adolescents (UP-A), is a transdiagnostic therapeutic intervention employing core dysfunction approaches, defined as such due to their attendance to features of various (emotional) disorders. The treatment may work to ameliorate symptoms more broadly by targeting cross-cutting features common to the range of disorders targeted. Specifically, the UP-A might lead to the successful treatment of an array of emotional disorders in youth by targeting processes common across these frequently co-occurring problems including poor distress tolerance, limited cognitive flexibility, and heightened avoidance.
  Arms: 16 Sessions of Therapeutic Intervention

SUMMARY:
The purpose of this protocol is to employ single case analytic strategies, including a multiple baseline design and novel modeling techniques to identify changes in cross-cutting features of emotional disorders as well as emotional disorder symptoms during the implementation of The Unified Protocol for the Treatment of Emotional Disorders in Adolescents (UP-A). The first aim is to investigate relationships between the use of UP-A treatment components and changes in measures of cross-cutting features of emotional disorders. The second aim is to investigate when and how reductions in symptoms of emotional disorders and presenting problems (i.e., symptoms of anxiety and depression, severity of presenting problems) occur throughout treatment.

DETAILED DESCRIPTION:
The goal of this study is to examine how a core dysfunction transdiagnostic psychotherapy for emotional disorders in youth influences change in cross-cutting features both theoretically linked to neuroticism and also targeted by this treatment. Another goal is to investigate change in symptoms of emotional disorders, including anxiety and depression, throughout the course of this treatment, the Unified Protocol for the Treatment of Emotional Disorders in Adolescents (UP-A).

My long-term goal is to identify ways to personalize an effective psychotherapy model for an array of youth emotional disorders by determining how and when implementation of different components of the UP-A influence change in mental health. My research objective in this study is to use group-level and novel single case analytic strategies to identify changes in emotional disorders during the implementation of the UP-A, a transdiagnostic form of cognitive behavior therapy (CBT) for adolescents. Specifically, I am interested in examining how features of the core dysfunction targeted by the UP-A, high neuroticism as well as symptoms of emotional disorders change throughout UP-A treatment. My central hypothesis is that adolescents with emotional disorders will display changes in measures of core dysfunction and reductions in symptoms of emotional disorders throughout UP-A treatment.

Aim 1: Investigate relationships between the use of UP-A treatment components and changes in measures of neuroticism, a core dysfunction that cuts across of emotional disorders. The main working hypothesis is that the administration of the UP-A will result in observable changes in measures of cross-cutting features of emotional disorders linked to neuroticism (cognitive flexibility, distress tolerance, and experiential avoidance). Such changes will occur after the introduction of relevant core principles of the UP-A. The proposed study is designed to determine whether change in these aspects of neuroticism and emotional disorder symptoms occur directly following the presentation of treatment components, or whether changes might instead be staggered throughout treatment.

Aim 2: Investigate when and how reductions in symptoms of emotional disorders (i.e., symptoms of anxiety and depression, severity of presenting problems) occur throughout treatment. Based on knowledge obtained from previous randomized, controlled trials (RCTs) focusing on the treatment of anxiety, depressive and related disorders, the main working hypothesis of Aim 2 is that the severity of emotional disorder symptoms will decrease from pre- to post-treatment.

Exploratory Aim 3: Investigate aspects of neuroticism as potential mechanisms of change in emotional disorder symptoms. The primary working hypothesis of Aim 3 is that changes in features of neuroticism targeted by the UP-A will precede changes in anxiety and depressive symptoms.

RESEARCH STRATEGY A. SIGNIFICANCE Anxiety, depression, and related emotional disorders are prevalent and impairing. They have high levels of symptom overlap and also share underlying temperament factors, including high neuroticism and low extroversion. The UP-A and similar core dysfunction-focused transdiagnostic therapy approaches may lead to successful treatment by targeting features that cut across emotional disorders.

B. INNOVATION Several studies of the UP-A indicate significant improvements in both anxiety and depression from pre- to post-treatment. Research foci have recently shifted in an effort to figure out why such these core-dysfunction treatments work. One step in this direction is determining whether cross-cutting features defining internalizing disorders (i.e., neuroticism and related constructs) might serve as mechanisms of treatment-based change in disorder symptoms and severity. One case study using the adult UP treatment found that changes in cross-cutting features, including mindfulness and cognitive reappraisal, changed prior to reductions in anxiety and depression. Within the child literature, a downward adaptation of the UP-A (as compared to anxiety-focused CBT program) demonstrated greater decreases in several cross-cutting features of emotional disorders, including sadness dysregulation and reappraisal, over the course of treatment. However, no study thus far has investigated change processes in cross-cutting features of emotional disorders, during treatment with the UP-A. The present study will advance our understanding of how implementation of the UP-A might lead to change in direct cognitive and behavioral targets as well as symptoms of emotional disorders in adolescents. An increased understanding of how, when and for whom the UP-A works is vital to personalizing this psychotherapy and maximizing its efficiency and uptake in future dissemination and implementation research. Another innovation of this investigation is its novel application of single-case research design methodology and modeling techniques in the analysis of time-sequence data. Although mechanisms of change may be investigated via large-scale RCTs of clinical interventions, the time, cost and labor of such trials can impede rapid dissemination efforts. This innovative single-case methodology allows clinical researchers to vet potential mechanisms of change more quickly to be used in future research.

C. APPROACH Research Design and Methods Overview. A non-concurrent multiple baseline design will be used. This type of design includes a series of A-B replications along with randomly assigned baseline periods (2, 3, or 4 weeks in this study; 3 participants per baseline condition). Repeated measures (adolescent- and parent-report of changes in cross-cutting features of emotional disorders and of disorder-specific symptoms) will be given weekly throughout treatment with more comprehensive assessment (adolescent- and parent-report as well as clinician-rated clinical severity and diagnostic impressions) occurring at pre- and post-treatment time points. The specific combination of analyses being used (nonparametric group-level comparisons to assess change at major time points [pre-, mid-, and post-treatment] as well as Simulation Modeling Analysis [SMA] to assess change over time in an individual) requires measures to be administered at a variety of time points (i.e., pre- and post- treatment, pre-, mid-, and post-treatment; weekly, respectively). Thus, change over time in weekly measures will be examined at pre-, mid-, and post-treatment at a group level, while change over time in weekly measures will be examined using weekly data (baseline, treatment repeated measures) at an individual subject level. Further, change over time in clinical interview data will be assessed from pre- to post-treatment.

Participants. A minimum of nine clinically anxious and/or depressed adolescents between the ages of 13 and 17 will be recruited via a university clinic, with at least three adolescents randomized to each baseline condition.

Intervention. Unified Protocol for the Treatment of Emotional Disorders in Adolescents (UP-A). Adolescents will complete 16 sessions of the Unified Protocol for the Treatment of Emotional Disorders in Adolescents in a fixed order. The UP-A is composed of 8 core modules, including Orienting to Treatment and Enhancing Motivation, Emotion Education, Introduction to Emotion-focused Behavioral Experiments, Awareness of Physical Sensations, Being Flexible in Your Thinking, Emotional Awareness, Situation-Based Emotion Exposures, Relapse Prevention.

Analytic Plan Data will be analyzed using a specific combination of analyses supported in the single case research design and clinical replication literature. Initial approaches will utilize data from weekly measures, plus those administered at pre-treatment, post-baseline, mid-treatment, and post-treatment time points. A second group of analyses, which will be used to measure change over time in variables of interest throughout treatment as well as potential mechanisms of treatment change, include the application of Parker and Hagan-Burke's (2007) clinical outcomes approach, which was established specifically for the analysis of single-case data as well as Simulation Modeling Analyses (SMA; [1-3, 30]), to identify changes in cross-cutting features and emotional disorder symptoms over the course of implementation of the UP-A.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents must be between 13 and 17 years of age
* Adolescents must have a primary DSM-5 anxiety or depressive disorder based on results of a diagnostic interview administered by a trained clinician at intake within protocol 20130139
* Adolescents must indicate elevated symptoms of depression via adolescent and/or parent report of symptoms (RCADS and/or RCADS-P Depression Subscale Index T-Score ≥ 60) and anxiety (RCADS and/or RCADS-P Total Anxiety Subscale Index T-Score ≥ 60) at intake
* If relevant, adolescents must be on a stable dose of any SSRI/SNRI medication
* Adolescents must self-report the ability to speak/read English sufficiently (and have at least one parent who can) to complete all study measures in English
* Adolescents must have a legal guardian available to sign study consents, remain present during assessments, and fill out study questionnaires.

Exclusion Criteria:

* Adolescents obtain a Full Scale IQ score below 80 on the Vocabulary and Matrix Reasoning subtests of an abbreviated IQ test
* Adolescents indicate possible cognitive delays that could interfere with successful completion of study procedures
* Adolescents currently receiving psychotherapy elsewhere.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2017-12-14 (Actual)

PRIMARY OUTCOMES:
Change in DSM-5 Anxiety and Depressive Disorder Diagnoses and Severity in Accordance with Anxiety Disorders Interview Schedule for the DSM-5, Child and Parent Versions (ADIS-5-C/P) | administered pre-baseline (prior to treatment initiation), post-baseline (after 2, 3, or 4 week waitlist period), and post-treatment (after 16 sessions of weekly treatment)
  measure of change in diagnostic severity of internalizing disorders pre- to post- treatment
Session to Session Change in a measure of emotion regulation in youth, Emotion Regulation Questionnaire-Child and Adolescent Form (ERQ-CA) | to be completed by adolescents weekly throughout baseline and treatment phases consisting of one assessment prior to initiating study, once weekly assessments during 2, 3, or 4 week baseline period, and assessments every week for 16 weeks
  measure of change in cognitive flexibility throughout baseline and treatment conditions
Session to Session Change in a measure of distress tolerance in youth, Distress Tolerance Scale (DTS) | to be completed by adolescents weekly throughout baseline and treatment phases consisting of one assessment prior to initiating study, once weekly assessments during 2, 3, or 4 week baseline period, and assessments every week for 16 weeks
  measure of change in distress tolerance throughout baseline and treatment conditions
Session to Session Change in a measure of avoidance behaviors in youth associated with emotional disorders, Emotional Avoidance Strategy Inventory for Adolescents (EASI-A) | to be completed by adolescents weekly throughout baseline and treatment phases consisting of one assessment prior to initiating study, once weekly assessments during 2, 3, or 4 week baseline period, and assessments every week for 16 weeks
  measure of change in experiential avoidance throughout baseline and treatment conditions
Session to Session Change in a measure of anxiety and depressive symptoms in youth (self-report), Revised Children's Anxiety and Depression Scale-Short Form (RCADS-Short Form) | to be completed by adolescents weekly throughout baseline and treatment phases consisting of one assessment prior to initiating study, once weekly assessments during 2, 3, or 4 week baseline period, and assessments every week for 16 weeks
  indicates change in levels of anxiety and depressive symptoms reported by adolescents throughout baseline and treatment conditions
Session to Session Change in a measure of anxiety and depressive symptoms in youth reported by parents, Revised Children's Anxiety and Depression Scale-Parent Report-Short Form (RCADS-P-Short Form) | to be completed by adolescents weekly throughout baseline and treatment phases consisting of one assessment prior to initiating study, once weekly assessments during 2, 3, or 4 week baseline period, and assessments every week for 16 weeks
  indicates change in levels of anxiety and depressive symptoms experienced by adolescents as reported by parents of adolescents throughout baseline and treatment conditions

SECONDARY OUTCOMES:
Session to Session Change in a measure of severity of presenting problems in youth, Top Problems | assessed weekly throughout the study (approximately 18-20 weeks)
  measure of change in adolescent-reported severity of presenting problems between sessions throughout treatment
Session to Session Change in Score on a measure of youth distress tolerance, The Behavioral Indicator of Resiliency to Distress (BIRD) | administered pre-baseline (prior to treatment initiation), at mid-treatment (after 7th session of weekly therapy), post-treatment (after 16 sessions of weekly treatment)
  secondary behavioral measure of between session change in distress tolerance throughout treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jill Ehrenreich-May, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ehrenreich-May J, Rosenfield D, Queen AH, Kennedy SM, Remmes CS, Barlow DH. An initial waitlist-controlled trial of the unified protocol for the treatment of emotional disorders in adolescents. J Anxiety Disord. 2017 Mar;46:46-55. doi: 10.1016/j.janxdis.2016.10.006. Epub 2016 Oct 17. PMID 27771133
- [Background] Farchione TJ, Fairholme CP, Ellard KK, Boisseau CL, Thompson-Hollands J, Carl JR, Gallagher MW, Barlow DH. Unified protocol for transdiagnostic treatment of emotional disorders: a randomized controlled trial. Behav Ther. 2012 Sep;43(3):666-78. doi: 10.1016/j.beth.2012.01.001. Epub 2012 Jan 18. PMID 22697453
- See also: Department of Psychology, Child and Adolescent Mood and Anxiety Treatment Program (currently recruiting study participants) — http://www.psy.miami.edu/camat/